CLINICAL TRIAL: NCT07381543
Title: A Prospective, Exploratory, Two-Arm Study of Adebrelimab Maintenance Therapy in Limited-Stage Small Cell Lung Cancer Following Either Induction Chemo-Adebrelimab Plus Concurrent Chemoradiotherapy or Concurrent Chemoradiotherapy Alone
Brief Title: Adebrelimab Maintenance Therapy for LS-SCLC Post Induction Chemo-Adebrelimab Plus CRT or CRT Alone
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Minglei Zhuo, Chief Physician, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ146
Record Dates: First submitted 2026-01-18; First posted 2026-02-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Localized Small Cell Lung Cancer
Keywords: Localized small cell lung cancer; Without prior systemic anticancer therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelimab Induction Therapy Group (Experimental): Induction Phase adebrelimab combined with etoposide and platinum-based chemotherapy Concurrent Chemoradiotherapy Phase Radiotherapy initiated prior to the third cycle of chemotherapy, no later than the start of the third cycle, combined with etoposide and platinum-based chemotherapy Maintenance Phase adebrelimab administered until disease progression, intolerable toxicity, or a maximum of 2 years of treatment.
  Interventions: Drug: Adebrelimab Induction Therapy Group
- Adebrelimab Maintenance Therapy Group (Experimental): Radiotherapy is initiated prior to the third cycle of chemotherapy, no later than the start of the third cycle, in combination with etoposide and platinum-based agents.
  Maintenance Phase adebrelimab is administered until disease progression, intolerable toxicity, or a maximum of 2 years of treatment.
  Interventions: Drug: Adebrelimab Maintenance Therapy Group

INTERVENTIONS:
Drug: Adebrelimab Induction Therapy Group — Induction Phase Adebrelimab: 1200 mg, intravenous infusion, every 3 weeks Etoposide: 100 mg/m², intravenous infusion, Days 1-3, every 3 weeks Platinum-based agent: Cisplatin 75 mg/m² or Carboplatin AUC 5, intravenous infusion on Day 1, every 3 weeks Radiotherapy: 45 Gy/30 fractions BID or 60-66 Gy/30 fractions QD.
  Maintenance Phase Adebrelimab: 1200 mg, intravenous infusion, every 3 weeks
  Arms: Adebrelimab Induction Therapy Group
Drug: Adebrelimab Maintenance Therapy Group — Concurrent chemoradiotherapy radiotherapy : 45 Gy/30 fractions BID or 60-66 Gy/30 fractions QD Etoposide: 100 mg/m², intravenous infusion, Days 1-3, every 3 weeks Platinum-based agent: Cisplatin 75 mg/m² or Carboplatin AUC 5, intravenous infusion on Day 1, every 3 weeks Maintenance therapy Adebrelimab: 1200 mg, intravenous infusion, every 3 weeks
  Arms: Adebrelimab Maintenance Therapy Group

SUMMARY:
Observation and Evaluation of the Efficacy and Safety of Adalimumab Combined with Chemotherapy Followed by Radiotherapy or Radiotherapy Alone as First-Line Treatment for Limited-Stage Small Cell Lung Cancer

DETAILED DESCRIPTION:
The study comprises two cohorts (A and B). Cohort A first receives two cycles of induction therapy combining PD-L1 inhibitors with chemotherapy, followed by two cycles of concurrent chemoradiotherapy and subsequent maintenance therapy with PD-L1 inhibitors. Cohort B first undergoes four cycles of concurrent chemoradiotherapy followed by maintenance therapy with PD-L1 inhibitors. Both cohorts continue treatment until disease progression or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old, male or female;
2. Patients with pathologically confirmed localized small cell lung cancer (as defined by the Veterans Administration Lung Study Group, VALG staging);
3. No anticipated need for tumor resection during the study period (including patients unsuitable for surgery or unwilling to undergo surgery);
4. No prior treatment for localized small cell lung cancer;
5. Presence of measurable tumor target lesions (meeting RECIST 1.1 criteria);
6. Expected survival > 3 months;
7. ECOG PS: 0-1;
8. Normal major organ function;

   1. Complete blood count (CBC) (without transfusion or hematopoietic growth factor correction within 14 days):

      Hemoglobin (Hb) ≥ 90 g/L; Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelet count (PLT) ≥ 100 × 10⁹/L; White blood cell count (WBC) ≥ 3.0 × 10⁹/L;
   2. Biochemical tests:

      Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (≤ 5×ULN for patients with liver metastases); Serum total bilirubin (TBIL) ≤ 1.5×ULN (≤ 3×ULN for subjects with Gilbert syndrome); Serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance ≥ 50 mL/min;
   3. Coagulation function:

      Activated partial thromboplastin time (APTT), International Normalized Ratio (INR), Prothrombin time (PT) ≤ 1.5×ULN;
   4. Doppler ultrasound assessment:

   Left ventricular ejection fraction (LVEF) ≥50%;
9. Women of childbearing potential must have a negative pregnancy test (βHCG) prior to treatment initiation. Women of childbearing potential and males (who have sexual intercourse with women of childbearing potential) must agree to use effective contraception continuously during treatment and for 6 months after the last dose.
10. Patients voluntarily participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Mixed SCLC and extensive-stage SCLC;
2. History of other malignancies within the past 5 years or concurrent malignancies, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, or superficial or non-invasive bladder cancer;
3. History of uncontrollable psychiatric disorders or severe intellectual or cognitive impairment;
4. Active, known, or suspected autoimmune disease; however, subjects with hypothyroidism requiring only hormone replacement therapy or skin conditions not requiring systemic treatment (e.g., vitiligo, psoriasis, or alopecia) are eligible;
5. Subjects with any severe and/or uncontrolled medical conditions, including:

   1. Subjects with uncontrolled blood pressure (systolic ≥150 mmHg or diastolic ≥100 mmHg);
   2. Subjects with ≥ Grade 2 myocardial ischemia or myocardial infarction, arrhythmias (including male QTc ≥ 450 ms or female QTc ≥ 470 ms), and ≥ Grade 2 congestive heart failure (New York Heart Association [NYHA] classification);
6. Severe unhealed wounds, ulcers, or fractures;
7. History of psychiatric drug abuse, alcoholism, or illicit drug use;
8. Active hepatitis (HBV reference: HBsAg positive with HBV DNA levels exceeding upper normal limit; HCV reference: HCV antibody positive with HCV viral load exceeding upper normal limit);
9. Human Immunodeficiency Virus (HIV, HIV 1/2 antibody) positive;
10. Patients unable to comply with the study protocol or participate in follow-up visits;
11. Patients deemed unsuitable for this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 3 years
  From subject enrollment to the first recorded disease progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
ORR | through study completion, an average of 3 years
  The proportion of subjects achieving complete response (CR) or partial response (PR) as their best overall response following treatment initiation, relative to the total number of subjects.
OS | through study completion, an average of 3 years
  Time from subject enrollment to death from any cause.
Adverse Events | From the first dose of durvalumab to 90 days after the last dose of durvalumab or start of subsequent anticancer treatment
  AEs that occurred from the first dose of durvalumab to 90 days after the last dose of durvalumab or start of subsequent anticancer treatment
DCR | through study completion, an average of 3 years
  The proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) as their best overall response following treatment initiation, relative to the total number of subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China